CLINICAL TRIAL: NCT00000647
Title: An Open Trial Combining Zidovudine, Interferon-alfa, and Recombinant CD4-IgG With Transplantation of Syngeneic Bone Marrow and Peripheral Blood Lymphocytes From Healthy gp160-Immunized Donors in the Treatment of Patients With HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: IRP 011; 11723 (Registry Identifier: DAIDS ES Registry Number); 90 I-0076; NIAID 90 CC-IRP011
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; IgG; Drug Evaluation; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Antigens, CD4; Zidovudine; Carrier Proteins; Interferon Type I
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — CD4 Immunoadhesins; Zidovudine; interferon alfa-n1; Bone Marrow Transplantation

INTERVENTIONS:
Drug: CD4-IgG
Drug: Zidovudine
Drug: Interferon alfa-n1
Procedure: Peripheral lymphocyte infusion
Procedure: Bone marrow transplant

SUMMARY:
To restore immunologic function and virus-free state in HIV-infected patients. Based on previous studies showing temporary improvement in immune function in HIV-infected patients using peripheral lymphocyte transfers and bone marrow transplantation, and based on studies documenting the antiretroviral effects of zidovudine (AZT) and interferon-alfa (IFN-A) as well as the preliminary test tube and patient studies suggesting anti-HIV effects of recombinant CD4-IgG, we propose to treat HIV-infected patients using combination antiretroviral therapy with transplantation of bone marrow and peripheral lymphocytes from previously immunized donors in an attempt to restore immunologic function and a virus-free state.

DETAILED DESCRIPTION:
Based on previous studies showing temporary improvement in immune function in HIV-infected patients using peripheral lymphocyte transfers and bone marrow transplantation, and based on studies documenting the antiretroviral effects of zidovudine (AZT) and interferon-alfa (IFN-A) as well as the preliminary test tube and patient studies suggesting anti-HIV effects of recombinant CD4-IgG, we propose to treat HIV-infected patients using combination antiretroviral therapy with transplantation of bone marrow and peripheral lymphocytes from previously immunized donors in an attempt to restore immunologic function and a virus-free state.

Three patients are treated with stable doses of AZT, IFN-A, and CD4-IgG for 12 weeks, followed by six peripheral lymphocyte infusions and transplantation of bone marrow from their respective identical twins. Following bone marrow transplantation, patients continue to receive the three drugs. Additional periods of lymphocyte apheresis and transfer may be offered to each donor/recipient pair.

ELIGIBILITY:
Inclusion Criteria

* Each patient must have an identical twin in a normal state of health with a normal screening lab panel and a normal immune profile who is documented to be antibody and culture and polymerase chain reaction (PCR) negative for HIV.
* Ability to provide informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malignancy other than Kaposi's sarcoma.

Patients with the following are excluded:

* Unwillingness to comply with current NIH Clinical Center guidelines concerning appropriate notification of all current sexual partners of an individual regarding his or her positive HIV serostatus and the risk of transmission of HIV infection.
* Presence of a serious opportunistic infection or other illness or condition that, in the opinion of the principal investigator, warrants exclusion from participation in the study.

Current use of illicit drugs or significant amounts of alcohol that, in the opinion of the principal investigator, would interfere with compliance with the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6
Dates: Study Completion 1994-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: KM Zunich, Study Chair
Locations (1):
- Natl Inst of Allergy & Infect Dis / Cln Ctr, Bethesda, Maryland, United States

REFERENCES:
- [Background] Zunich KM, Easter M, Owen C, Walker R, Davey R, Wilson W, Leitman S, Fauci AS, Lane HC. Bone marrow transplantation and adoptive transfer of peripheral blood lymphocytes from gp160-immunized syngeneic donors combined with zidovudine, interferon-alpha, and recombinant CD4-IgG in the treatment of HIV infection. Int Conf AIDS. 1991 Jun 16-21;7(2):77 (abstract no THB82)